# **Clinical Investigational Plan**

# **DINR**

| Full title of Investigation: | Digital Interventions in Neuro-Rehabilitation: A digital neuro intervention (DNI) for word retrieval. A small scale randomised clinical trial to test a web-based therapy application for people with naming difficulties with mild- moderate Dementia (Gotcha!). |
|---|---|
| Short title: | Digital Interventions in Neuro-Rehabilitation (DINR):<br>Gotcha! |
| Version and date of Clinical Investigation Plan (CIP): | Version 6.0, 15.01.2024 |
| Sponsor: | University College London (UCL) |
| Sponsor CIP number: | 18/0071 |
| Funder (s): | NIHR |

## **Revision History:**

| Version numbers | Date | Summary of revisions in the case of amendments | Protocol Updated by |
|---|---|---|---|
| 1 | 18.03.2018 | | |
| 2 | 31.07.2018 | | Henry Coley-Fisher Dr. Catherine Doogan |
| 3 | 07.02.2019 | Separating both apps | Dr Catherine Doogan<br>Emily Upton |
| 4 | 25.02.2019 | Statistical recommendations from MHRA added. | Henry Coley-Fisher<br>Alex Leff |
| 5 | 15.03.2019 | Sample size amended | Emily Upton |
| 6 | 15.01.2024 | Clarification added to the Inclusion criteria that mild/moderate dementia, includes AD/vascular and mixed, primary progressive aphasia, and dementia with Lewy bodies | Aygun Badalova |

## **Signatures**

The Chief Investigator (CI) and the JRO have discussed this Clinical Investigation Plan (CIP). The investigator agrees to perform the investigations and to abide by this CIP.

The investigator agrees to conduct the Investigation in compliance with the approved CIP, EU Good Clinical Practice (GCP) and UK Regulations for Devices (SI 2002/618; as amended) for regulated studies, the UK Data Protection Act (2018), the Trust Information Governance Policy (or other local equivalent), the Research Governance Framework (2005 2<sup>nd</sup> Edition; as amended), the Sponsor's SOPs, and other regulatory requirements as amended.

| Chief investigator | | |
|-------------------------------|-----------|------|
| Prof Alex Leff | | |
| | Signature | Date |
| <b>Sponsor Representative</b> | | |

## **Contents**

| Sponsor | 7 |
|---|---|
| Principal Investigator, Coordinating Investigator and Investigation site(s) | 7 |
| A.1 Overall Synopsis of Clinical Investigation | 8 |
| Inclusion criteria | |
| b) Exclusion criteria | |
| No diagnosis of developmental language disorders | |
| A.2 Background and Rationale | |
| A.3 Identification and description of the Investigational Device | |
| • | |
| A.4 Justification for the design of the clinical investigation | 13 |
| A.5 Risks and benefits of the Investigational device and clinical Investigation | 14 |
| A.6 Objectives and hypotheses of the clinical investigation | 15 |
| A6.1 Hypotheses | |
| A6.2 Primary Objective | 15 |
| A6.3 Secondary Objective(s) | 15 |
| A.7 Design of the clinical investigation | |
| A.7.1 General | |
| A.7.2 Investigational device and comparators | |
| A.7.3 Subjects | |
| a) Inclusion criteria | |
| b) Exclusion criteria | |
| No diagnosis of developmental language disorders | |
| c) Criteria and procedures for subject withdrawal or discontinuation | |
| d) Point of enrolment | |
| e) Total expected duration of the clinical investigation | |
| f) Expected duration of each subject's participation | |
| g) Number of subjects included in the clinical investigation | |
| h) Estimated time needed to select this number (i.e. enrolment period) | |
| Subject Eligibility | |
| A7.5 Recruitment | |
| A7.5 Randomisation Procedures | |
| A.7.6 Procedures | 20 |
| A.8 Informed Consent Process | 20 |
| Procedure of gaining consent | 21 |
| A.9 Schedule of assessments and interventions by visit | 21 |
| A.10 Device accountability | 23 |
| A.11 Monitoring Plan | 23 |
| a. Confidentiality | 23 |
| b. Record keeping and archiving | 23 |
| A.13 Data Management | |
| A13.1 Procedures for data review, database cleaning, and issuing and resolving data queries | |
| A13.2 Procedures for verification, validation and securing of electronic clinical data systems | |
| A13.3 Data retention | |
| A13.4 Clinical quality assurance | |
| A13 5 Completion of Case Report Forms | 27 |

| A13.6 Review and Return of Completed Documentation | 28 |
|---|---|
| A13.7 Retention of Documentation | |
| A13.8 Training | 29 |
| A.14 Amendments to the CIP | 29 |
| A.15 Deviations from clinical investigation plan | 29 |
| A.15.1 Procedures for recording, reporting and analysing CIP deviations | 29 |
| A.15.2 Procedure for reporting any protocol deviations | |
| The clinical investigation shall not commence recruitment until all REC, regulatory (if applicable) an | |
| permission) is received. All additional requirements imposed by the REC or regulatory authority will | |
| A.17 Insurance | |
| A.18 Adverse events, adverse device effects and device deficiencies | 31 |
| a-c) Definitions | 31 |
| An adverse event does not include: | |
| d) Reporting requirements and timelines | |
| e) Assessments of adverse events | |
| Seriousness | |
| Causality | |
| Expectedness | |
| f) Procedures for recording and reporting Adverse Events and Device Deficiencies | 35 |
| Investigator responsibilities: | |
| Reporting of all Adverse Events and Device Deficiencies: Investigator and Sponsor responsib | |
| Progress reports | |
| a) Anticipated adverse events and adverse device effects (ADEs), together with their likely incide mitigation or treatment. | , |
| A.19 Oversight Committees | |
| A.20 Vulnerable population | 39 |
| A.21 Suspension or premature termination of the clinical investigation | |
| A21.1 Subject Withdrawals and Discontinuation | 40 |
| A.22 Definition of End of Trial | |
| A.23 Publication policy | 41 |
| A 24 Rihliogranhy | 43 |

## LIST OF ABBREVIATIONS

| ADE | Adverse Device Effect |
|---------|-----------------------------------------------------|
| AE | Adverse Event |
| CA | Competent Authority |
| CI | Chief Investigator |
| CIA | Clinical Investigation Agreement |
| CIP | Clinical Investigation Plan |
| CRF | Case Report Form |
| CRO | Contract Research Organisation |
| DINR | Digital interventions in Neuro-rehabilitation |
| DNI | Digital Neuro-intervention |
| DCF | Data Clarification Form |
| DD | Device Deficiency |
| EC | European Commission |
| EU | European Union |
| EUDAMED | European Medical Devices Regulatory Database |
| G! | Gotcha! |
| G!m | Gotcha! Maintenance |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HRA | Health Research Authority |
| IB | Investigator Brochure |
| ICF | Informed Consent Form |
| IMD | Investigational Medical Device |
| ISF | Investigator Site File |
| JRO | Joint Research Office |
| MA | Marketing Authorisation |
| MHRA | Medicines and Healthcare products Regulatory Agency |
| NCA | National Competent Authority |
| NHS | National Health Service |
| NHS R&D | National Health Service Research & Development |
| NICE | National Institute of Clinical Excellence |
| NIHR | National Institute of Health Research |
| NIST | National Institute of Standards and Technology |

| PI | Principal Investigator |
|-------|---------------------------------------------|
| PIS | Participant Information Sheet |
| QA | Quality Assurance |
| QC | Quality Control |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SALT | Speech and Language Therapy |
| SOP | Standard Operating Procedure |
| TMG | Trial Management Group |
| UADE | Unanticipated Adverse Device Effect |
| UK | United Kingdom |
| USADE | Unanticipated Serious Adverse Device Effect |
| WTCN | Wellcome Trust Centre for Neuroimaging |

## **Sponsor**

| Sponsor's representative | UCL/UCLH Joint Research Office, |
|--------------------------|---------------------------------|
| Samim Patel | 4 <sup>th</sup> Floor West, |
| | 250 Euston Road, |
| | London NW1 2PG |
| | Email: samim.patel@ucl.ac.uk |
| | Tel: 0207 679 9320 |

# Principal Investigator, Coordinating Investigator and Investigation site(s)

| Chief Investigator (CI)<br>Professor of Neurology | Prof Alex Leff,17-19 Alexandra House, Queen Square, WC1N 3AZ <a href="mailto:a.leff@ucl.ac.uk">a.leff@ucl.ac.uk</a> |
|---|---|
| | 0207 279 1129 |
| Principal Investigator (PI) | Prof Alex Leff,17-19 Alexandra House, Queen Square, WC1N 3AZ |
| Professor of Cognitive Neurology | a.leff@ucl.ac.uk |
| & Honorary Consultant Neurologist | 0207 279 1129 |
| Co-Investigator | Dr. Catherine Doogan, UCL, <u>c.doogan@ucl.ac.uk</u> , (Clinical Psychologist) |
| | Dr. Jennifer Crinion, UCL, <u>j.crinion@ucl.ac.uk</u> (Speech and Language therapist) |
| | Aygun Badalova, aygun.badalova.20@ucl.ac.uk, Research Assistant, NeurotherapeuticsLab |
| | ICN 17-19 Queen |
| | Square, London, |
| | WC1N 3AZ |
| | 0207 279 1134 |
| Add in other involved investigators | Wellcome Centre for Human Neuroimaging (WCHN), Institute of |
| as required | Neurology, UCL |
| | Head of Center Prof Cathy Price. |
| Statistician | Dr Tom Hope, |
| | Senior Research Associate |
| | Wellcome Centre for Human Neuroimaging |
| | University College London |
| | London WC1N 3AR |

### A.1 Overall Synopsis of Clinical Investigation

**Title:** Digital Interventions in Neuro-Rehabilitation (DINR): A digital neuro intervention

(DNI) for word retrieval (anomia). The development and testing of a web-based therapy application for people with naming difficulties who have mild- moderate

Dementia (Gotcha!).

Short title: Digital Interventions in Neuro-Rehabilitation (DINR): Gotcha!

**Device:** A digital intervention in Neuro-rehab (DNI). A word-retrieval app for people who have

mild-moderate Dementia.

**Objectives:** Digital Interventions in Neuro-Rehabilitation (DINR): A digital neuro intervention

(DNI) for word retrieval.

**Gotcha!** will be for people with dementia who have difficulty naming people they

know well.

The main objective is to ascertain if Gotcha! improves naming performance on trained

items?

Secondary outcomes will include improvements in social activity and participation

and participant and/or carer reported outcome measures (PROMS).

We also plan to capture brain-based data (functional and structural MRI and MEG)

in order to test a series of secondary hypotheses relating to both how and why the

therapy may work in some participants but not in others.

**Type of Investigation:** A single-site randomised control trial.

Investigation design and methods:

This is a summary of the protocol for the study funded by the National Institute of Health Research (NIHR). The main aim of this Phase 2 study is to test the clinical efficacy of the DNI through a randomised small-scale clinical trial. The participants will take the app home on a mobile device and 'play' the therapy. After the trial the participant will return the device and we will delete any content on the device and

reload the DNI.

Gotcha!: Gotcha! is a structured small scale clinical trial. Participants will be

randomised into two groups: either Gotcha! (therapy only) or Gotcha! maintenance.

Participants will complete 7 assessment sessions (T1-T7) at UCL, they will complete neuropsychological assessments, receive brain imaging scans and complete a program of therapy using the DNI. One group will complete a maintenance period after the initial therapy block.

20 control participants will be recruited in the Gotcha! study to generate a range of normality on our non-standardised tests. The control participants will be invited to one testing session at the Institute of Cognitive Neuroscience where they will complete behavioural tests and have two brain scans (1 MEG and 1 MRI).

Investigation duration per participant:

54 weeks

Estimated total Investigation duration:

3 years

Planned Investigation sites:

Single-site is **UCL**.

Total number of participants planned:

**44**: 44 Participants with AD/vascular and mixed, primary progressive aphasia, and dementia with Lewy bodies

Main inclusion/exclusion criteria:

Inclusion criteria

Person with mild/moderate dementia, including AD/vascular and mixed, primary progressive aphasia, and dementia with Lewy bodies

Self-reported proper naming difficulty which we will then assess at Time Point 1

English as their dominant language

Able to tolerate MRI brain scan

Able to give informed consent

Able to use the DNI (app)

b) Exclusion criteria

No diagnosis of developmental language disorders

No diagnosis of severe dementia or primary progressive aphasia

No major co-existing neurological or psychiatric diagnosis

No contraindications to brain scanner (e.g. the presence of ferromagnetic implants or other metallic or electronic objects in the body, weight over 24

stone, claustrophobia or pregnancy).

Behavioural data:

Statistical

methodology and

analysis:

Behavioral baseline data will be analysed using minimisation (Altman, BMJ 2005) to ensure that the two groups are not unbalanced on key demographic variables, including

baseline performance during the randomisation procedure.

Data from all time points will be analysed using a repeated-measures ANOVA to determine whether there is an interaction between time (therapy block vs baseline) and item (trained vs untrained). The effect of the between-group factor (therapy type) is a secondary outcome measure which will also be analysed using a repeated measure

secondary successive measure which will also be analysed using a repeated measure

ANOVA but with this extra factor added in: more formally, a three-way interaction

between time (therapy block vs baseline), item (trained vs untrained) and therapy type

(Gotcha! vs Gotcha! maintenance).

Neuroimaging data:

Collected at three of the time points. Structural magnetic resonance imaging (MRI)

data will be used to identify the lesion location and to aid co-registration of the

functional MEG data. Brain structure at the three time points will be analysed using

Voxel-Based Morphometry (Ashburner and Friston 2000) within the Statistical

Parametric Mapping software (SPM12) to identify whether these therapies induce any

structure brain changes over time. We will employ multi- parameter mapping MRI

methodology for the structural brain scans (Callaghan et al, 2014).


A.2 Background and Rationale

**Background** 

The number of people with dementia in the UK is forecast to increase by 40% over the next 12 years and 156%

over the next 38 years (Prince et al., 2014). People with all stages of Alzheimer's disease (AD) report forgetting

even very familiar people's names, which patients find annoying and embarrassing (Werner, 2004). This

therapy speaks to the James Lind Alliance's dementia top priority, "What are the most effective components of

care that keep a person with dementia as independent as they can be at all stages of the disease in all care

settings?" Several case studies and one group study have shown that patients with AD can significantly improve

proper name recall with training; the effects last months after training is completed (Clare et al., 2002). Given

the prevalence of mobile phone technology with inbuilt cameras and the rapid rise in usage in the 64-74 year old

bracket, we will develop a name-training intervention that allows people with proper name recall impairments to

take pictures of and add the name of people that they wish to name. The app will include voice recognition

software so that our bespoke adaptive algorithm (developed with Prof Mark Huckvale at UCL) will be able to

adaptively cue users depending on their speech output.

Gotcha! will provide an app-based therapy for people with dementia who have difficulty naming people they

know well.

This Digital Neuro Intervention (DNI) will provide the opportunity for the necessary increased rehabilitation to

help people recover lost naming function. This will alleviate NHS Speech and Language Therapist (SALT) time

and put users in control of when and where they carry out practice-based language therapy.

A.3 Identification and description of the Investigational Device

**Purpose** 

Gotcha! will provide an app-based therapy for people with dementia who have difficulty naming people they

know well.

What does it do?

The therapy element works via mass practice and feedback to the users on a trial-by-trial basis. The DNI is very

simple in a way; it just presents a long series of pictures for users to name. This DNI will use speech recognition

(SR) software in order to make a binary decision as to whether the user said the correct word or not. This affects

what the next trial (object to name) is and what auditory cue (if any) is provided the next time the user has to name

the same item.

\*The speech will be recorded on the device but no other identifiable information will be stored on it. When the participant finishes the trial, we will delete all information on the device.

## What is the clinical trial design?

A small, well-defined sample of patients with the potential to benefit from the DNI will be recruited. The main outcome measure is whether the DNI is effective at improving naming impairments. This comparison is within-subject and is achieved by comparing post-therapy measures to multiple baseline measures. We are also comparing two different versions of the therapy (a between group comparison) to answer our secondary question of whether the therapy can be optimised. Outcome measures will be collected by the research team using a variety of standardized and non-standardized tests of language and cognition.

The DNI will be introduced to the participant when attending a testing session. One of the research team will explain how to use the DNI, provide instructions for the user, and give some time for practice items. When confident that the participant can use the DNI independently, the participant will take the device home and continue their therapy (suggested therapy time is 5-10 hours per week) which will be simultaneously monitored by the research team. The research team will also check in on the participant weekly to trouble shoot any difficulties they may have (whether motivational or technical). When the participant has completed the therapy block, we will invite them in again for testing and they will return the mobile device with the DNI on it. The participants who continue to receive standard care during the therapy block will be asked to record and submit details to the research team.

### A.4 Justification for the design of the clinical investigation

## Why is the research considered worth doing?

Standard (face to face) Speech and Language Therapy (SALT) has a huge evidence-base but patients in the NHS have unmet therapy needs due to a lack of resources. The evidence from speech-therapy highlights the amount of time-on-task required to improve patients' ability to communicate. Naming problems are common and impact on the patients' wellbeing and social inclusion. There is also good evidence that current existing therapeutic approaches work.

In the NHS a patient with Alzheimer's Dementia are likely to receive little or no SALT. Our solution to the lack of available SALT therapy is to produce digital neuro-interventions that give patients the opportunity to practice scientifically validated, impairment based therapy when and where it suits them which gives them access to optimum therapy dose.

We know that therapy is effortful for patients who can sometimes be too fatigued when the therapist comes to do their session. This digital neuro-intervention will provide optimum availability of therapy and therefore place the patient in control of how much they do. However, as we recognise it is still effortful we hope to make the therapy engaging through adaptive and exciting software. The adaptiveness will serve to reward the patients for their efforts without ever making them feel like they are failing. This will hopefully boost how long they spend in therapy and therefore make greater gains.

There are therapy apps available for patients but the scientific basis for them is lacking and none are targeted for proper name anomia. By using speech recognition software our intervention will be uniquely designed to be used by patients with word retrieval impairments.

## What new information will the research provide?

The concept of the therapy component is based on standard SALT practice and thus has a strong proof of concept basis, as do our proposed outcome measures. The novel component is packaging it in a user- friendly web-app that is designed for and by people with word-retrieval problems. We will test the efficacy in a randomized-controlled trial (Phase 2). These digital neuro-interventions will be in contrast to the plethora of apps available online claiming cognitive training without having scientific proof.

The Gotcha! research study is a small-scale, randomised clinical trial for participants with mild to moderate dementia who have difficulty naming the people they know well (proper name anomia). The main research question is whether Gotcha! therapy improves participants' ability to freely name the people they know well. We will test this hypothesis by assessing participants' naming abilities on two matched lists of people, half are trained and half remain untrained.

A secondary question relates to maintenance of therapy gains, we will test this hypothesis by creating two different versions of Gotcha!, 'standard Gotcha!' and 'Gotcha! Maintenance'. These two versions are identical for the first block of therapy but differ thereafter in that the maintenance version continues to top up participants with brief training sessions over the next block while those in the standard group do not have any further interactions with the therapy. Participants will be randomised (using minimisation) to one of the two versions of the therapy. The main outcome measure will be a clinically relevant improvement on the naming ability of the trained items (compared to untrained control items). Secondary outcomes will include improvements in social activity and participation and participant and/or carer reported outcome measures (PROMS).

We also plan to capture brain-based data (functional and structural MRI and MEG) in order to test a series of secondary hypotheses relating to both how and why the therapy may work in some participants but not others. All brain imaging will be outside of standard care for the participants and take place at UCL by trained staff.

Digital Interventions in Neuro-Rehabilitation: Gotcha! CIP. Version: 6, Date: 15.01.24, IRAS #: 237795


## A.5 Risks and benefits of the Investigational device and clinical Investigation

The potential clinical benefit to the participants is that they will be receiving more therapy through the DNI that they could ever receive from the NHS. This in turn will provide opportunity for them to improve their word retrieval which can be a distressing impairment.

A full risk assessment and mitigation plan for each risk relating to the investigational device and the clinical investigation is detailed in a separate document entitled: Risk Assessment CTIMP Gotcha!.

The table below summaries the risks and mitigations of all tests above standard care that are being performed:

Table 1

| Intervention | Potential risk | Risk Management |
|---|---|---|
| MRI | Only if any contraindications are missed or not reported. | Performed by trained member of staff. |
| | These contraindications may include the presence of any metal in the body. | Follow trust standard operational procedures by obtaining surgical history of exposure to metal, metallic dental work and other potential MRI contraindications. |
| | Discomfort or anxiety in the MRI scanner may occur due to the noise and enclosed space. | These potential risks will be reduced by providing an alarm bulb in the case of any uncertainty discomfort, or distress. Noise from the scanner will be attenuated by the use of earplugs and noise-shielding headphones |
| X-Ray | Exposure to ionising radiation | Performed by trained member of staff. Following trust protocols. The standard dose is equivalent to ~0.005% of average annual radiation dose in the UK |

The classification of medical devices in the European Union is outlined in Annex IX of the Council Directive 93/42/EEC (as amended). There are four classes, ranging from low risk to high risk.

Class I

Class IIa

Class IIb

Class III

The Medical Device used in this investigation is classified as Class IIa

A.6 Objectives and hypotheses of the clinical investigation

A6.1 Hypotheses

**H1-Primary:** 

Does Gotcha! improve naming performance on trained items?

This is a within-subject comparison. The criteria for success is a 10% (raw, or unstandardized) relative

improvement in performance. This effect size was used in the recent Big Cactus study.

**H2-Secondary:** 

Does Gotcha! maintenance keep participants at their maximum achieved level compared to standard Gotcha?

This is two factor analysis with both a within-subject factor (trained vs. untrained items) and a between-group

factor (Gotcha! maintenance vs. standard Gotcha). The criteria for success is a 10% (raw, or unstandardized)

relative difference in performance. This effect size was used in the recent Big Cactus study.

A6.2 Primary Objective

Does Gotcha! improve naming performance on trained items?

A6.3 Secondary Objective(s)

We believe that using this DNI will improve word retrieval on trained items by providing a known therapy used by

SLT's through a digital app and by enabling an increased dose of therapy. However, we also believe that by using

this DNI and practicing every day, there will be changes in participants' brain structure and in the health of the

participants and their carers.

• Does Gotcha! maintenance keep participants at their maximum achieved level compared to

standard Gotcha?

• Are the therapy effects item-specific or do we see generalization to untrained items?

• Are the effects of the DNI therapy limited to the language domain alone or do they improve in

other cognitive domains (e.g. sustained attention)?

• Does the DNI improve participant's social activity and participation?

• Is the DNI acceptable to participants (can they use it easily)?

- Is the DNI acceptable to participants' carers?
- Does the DNI improve carer health/well-being?
- Does the DNI have any economic benefits?
- Can baseline structural brain imaging explain participants' responses to the DNI?
- Can baseline structural brain imaging be used to predict incoming participants' response to the DNI?
- Can repeated-measures structural or functional brain imaging identify participant's brain areas that change in response to the DNI?

## A.7 Design of the clinical investigation

### A.7.1 General

Gotcha! is a small scale, randomised, clinical trial for participants with word retrieval impairments who have Dementia. Participants (with AD) will be randomised into two groups: either Gotcha! (6 weeks of therapy only) or Gotcha! maintenance: 6 weeks of therapy plus a further 12 weeks of 'top-up' therapy to maintain gains).



The naming tests will be audio recorded. Nothing will be video recorded.

### **Control Participants**

Digital Interventions in Neuro-Rehabilitation: Gotcha! CIP. Version: 6, Date: 15.01.24, IRAS #: 237795 

20 control participants will be recruited in the Gotcha! study to generate a range of normality on our non-standardised tests. The control participants will be invited to one testing session at the Institute of Cognitive

Neuroscience where they will complete behavioural tests and have two brain scans (1 MEG and 1 MRI).

A.7.2 Investigational device and comparators

The device which the DNI will be uploaded onto will be stored in a secure cabinet in the ICN building. After the

trial ends, the DNI will be deleted from the app and the mobile devices will be stored or used by Prof Leff as he

sees fit. No data will remain on the individual devices.

A.7.3 Subjects

a) Inclusion criteria

Person with mild/moderate dementia, including AD/vascular and mixed, primary progressive aphasia, and

dementia with Lewy bodies

Self-reported proper naming difficulty which we will then assess at Time Point 1

English as their dominant language

Able to tolerate MRI brain scan

Able to give informed consent

b) Exclusion criteria

No diagnosis of developmental language disorders

No diagnosis of severe dementia or primary progressive aphasia

No major co-existing neurological or psychiatric diagnosis

No contraindications to brain scanner (Phase 2 only e.g. the presence of ferromagnetic implants or

other metallic or electronic objects in the body, weight over 24 stone, claustrophobia or pregnancy).

## c) Criteria and procedures for subject withdrawal or discontinuation

A participant may be withdrawn from the trial whenever continued participation is no longer in the participant's best interests, but the reasons for doing so must be recorded. Reasons for discontinuing the trial may include:

- Disease progression whilst in the study
- Intercurrent illness
- Patients withdrawing consent
- Persistent non-compliance to protocol requirements.

### d) Point of enrolment.

Participants are enrolled at T1 (first time point) as this is where consent is obtained. They are randomized at T3 (after all three baseline measurements have been collected).

## e) Total expected duration of the clinical investigation

3 years.

### f) Expected duration of each subject's participation

54 weeks (patients with AD only)

### g) Number of subjects included in the clinical investigation

44

### h) Estimated time needed to select this number (i.e. enrolment period)

2.5 years

#### **Subject Eligibility**

Once written informed consent has been obtained, the Case Report Form will be completed to document adherence to the inclusion and exclusion criteria.

Where a subject fails to fulfil any element of the inclusion and exclusion criteria, this will be documented and the signed consent form and completed inclusion/exclusion criteria will be retained by the Principal Investigator. The subject will not advance any further into this clinical investigation.

## **Subject Identification**

When a subject is identified and considered eligible for entry into this clinical investigation, the subject will be

allocated the next available investigation number (subject ID number).

For subjects enrolled, this number will consist of 01 for the first subject, 02 for the second subject and so on. This

number will be the unique identifier of the subject and written on each page of the paper/electronic Case Report

Form booklet and all other documentation relating to that subject.

Each subject that is enrolled into the study will have their study participation recorded and details of the device

recorded in their hospital notes. A copy of their signed consent form and patient information sheet should also be

placed on his/her hospitals notes to identify the subject as participating in a Clinical Investigation.

A7.4 Recruitment

Participant recruitment at a site will only commence when the trial has been initiated by the Sponsor (or it's

delegated representative), and issued with the 'Open to Recruitment' letter.

Suitable participants will be identified by the clinical care teams in two NHS patient identification centres

(CANDI and NELFT) and advertised in their centre. When consented to be contacted about participation in

research, participants will be contacted by telephone by a member of the research team (usually Dr Doogan or a

research assistant but may include other members of the team). We may also advertise in local community

groups e.g. Alzheimer's Society.

The basic details of our study will be publicised on other appropriate websites and social media.

A7.5 Randomisation Procedures

After consent has been gained and the participants have completed 3 sessions of baseline testing, the CI will

randomise the participants using minimisation. This will determine which version of the therapy the participant

will use: Gotcha! only or Gotcha! maintenance groups.

Participants are considered to be enrolled into the trial following: consent, pre-treatment assessments, confirmation

of eligibility, allocation of the participant trial number and treatment by the central coordinating team/remote

system. The completion of the randomisation process happens at time point 3 and so they will have been enrolled

since Time point 1.

Digital Interventions in Neuro-Rehabilitation: Gotcha! CIP. Version: 6, Date: 15.01.24, IRAS #: 237795


### A.7.6 Procedures

The DNI will be introduced to the participant when attending a testing session. One of the research team will explain how to use the DNI, provide instructions for the user, and give some time for practice items. When confident that the participant can use the DNI independently, the participant will take the device home and continue their therapy (suggested therapy time is 5-10 hours per week) which will be simultaneously monitored by the research team. The research team will also check in on the participant weekly to trouble shoot any difficulties they may have (whether motivational or technical). When the participant has completed the therapy block, we will invite them in again for testing and they will return the mobile device with the DNI on it. The participants who continue to receive standard care during the therapy block will be asked to record and submit details to the research team.

Brain Imaging will also take place. This will happen 3 times, at time-points 2, 3 and 4. The scans will take place in UCL, carried out by trained staff, on the same day as the participants are coming in for behavioural testing and will last approximately 30 minutes.

#### A.8 Informed Consent Process

We understand it is the responsibility of the Investigator, or a person delegated by the Investigator, to obtain written informed consent from each subject prior to participation in the Investigation, following adequate explanation of the aims, methods, anticipated benefits and potential hazards of the study.

The person taking consent will be GCP trained, suitably qualified and experienced, and have been delegated this duty by the CI/PI on the delegation log.

A week will be given for consideration by the patient before taking part. The PI must record when the patient information sheet (PIS) has been given to the patient. [If the amount of time between the PIS being given and the date of consent are less than 24 hours, the PI will explain the rationale for this]. It must be recorded in the medical notes when the participant information sheet (PIS) has been given to the participant.

The Investigator or designee will explain the patients are under no obligation to enter the Investigation and that they can withdraw at any time during the Investigation, without having to give a reason.

No clinical Investigation procedures will be conducted prior to taking consent from the participant. Consent will not denote enrolment into Investigation. A copy of the signed Informed Consent Document will be given to the participant. The original signed form will be retained at the study site and a copy placed in the medical notes.

If new safety information results in significant changes in the risk/benefit assessment, the consent form will be reviewed and updated if necessary and subjects will be re-consented as appropriate

The procedures for consent outlined in the Standard Operating Procedure for informed consent form (UCL) will be adhered to. A written record of the checks made for competence to consent will be kept along with other information in each patient's Case Report Form. The CI will also ensure that written consent is witnessed, preferably by a relation or carer of the patient, or if not, by an independent witness present at the Welcome Trust Centre for Neuroimaging, UCL (WTCN).

Written, informed consent will be obtained for all participants. We plan to follow published guidelines for addressing consent issues in aphasic patients (Penn, Frankel et al. 2009).

Only members of the clinical care team will be identifying and approaching patients.

The research team has considerable experience of working with patients with impaired speech and language abilities (there are four speech and language therapists on the team), and will take the required time and attention to ensure that the requirements and risks of the study are thoroughly understood (by both the participant and, where appropriate, a family member or carer) before consent is obtained.

## Procedure of gaining consent

The clinical teams in the CANDI and NELFT PICs will identify potential participants and obtain consent to be contacted by the research team to discuss the Gotcha! study in more detail. Written and visual information materials will be distributed where required.

Potential participants will be telephoned again at least 1 week after initial contact, by Dr Doogan or the research assistant to answer any further questions and, if appropriate, to arrange the first testing appointment at the participating site. When participants come into their first testing appointment, written consent will be obtained.

At the first and subsequent appointments, potential participants will have a further opportunity to ask questions about the study.

If there is any change in capacity as indicated by a carer, the participant or a member of the research team, Dr Doogan, a Clinical Psychologist, will assess this and discontinue if found to be changed.

## A.9 Schedule of assessments and interventions by visit

| Time-<br>point | Gotcha! |
|---|---|
| <b>T1</b> | Baseline neuropsychological testing |
| | Addenbrooke's cognitive Examination (ACE-III) |
| | Self-report and carer-report outcome measure |
| | • Language testing |
| <b>T2</b> | Self-report and carer-report outcome measures |
| | Language and cognitive testing |
| | Brain Imaging |
| Т3 | Self-report and carer-report outcome measures |
| | Brain imaging |
| | Language and cognitive testing |
| | Participants are randomised to either Gotcha! or Gotcha! Maintenance groups |
| | Participants receive a mobile device with the DNI on it.Both groups start therapy intervention. |
| T4 | Self-report and carer-report outcome measures |
| | Brain Imaging |
| | Language and cognitive testing |
| | Participants in the standard Gotcha! block no longer get the therapy and maintenance group begins to receive maintenance therapy. |
| T5 | • ACE-III |
| | • Self-report and carer-report outcome measures. |
| | Language and cognitive testing |
| | G!m group stop maintenance therapy. |
| | The mobile device with the DNI is taken away. |
| Т6 | Self-report and carer-report outcome measures |
| | Language and cognitive testing |
| <b>T7</b> | Self-report and carer-report outcome measures. |
| | • ACE-III |
| | Language and cognitive testing |

Some assessments may be audio and video recorded to ensure accuracy when scoring.

We will inform participants' GPs and therapists (if they have one) of their involvement in the study.

A.10 Device accountability

The DNI (software) will be given to each participant to use on hardware (a tablet computer) purchased from the

grant and thus belonging to UCL. Because the software uploads data periodically to the database (on the UCL

secure virtual server), we are able to tell when participants are using it. At the end of the trial block, the DNI (and

tablet computer) are passed back to the research team and will be recycled for a future participant to use.

**A.11 Monitoring Plan** 

Case Report Forms (CRFs) will be completed by the investigator and/or his/her delegates at each timepoint. These

will record any potential AEs or ADEs. These data will be collated and passed onto the IDMC for their view on

safety. As each participant has several timepoints when they are not using the DNIs, we will be able to perform

within-subject analyses for the IDMC to see if rates of AEs or ADEs are higher in the DNI therapy blocks.

a. Confidentiality

All data will be handled in accordance with the UK Data Protection Act 1998. The CRFs will not bear the subject's

name or other personal identifiable data. The subject's Investigation identification number, will be used for

identification. Subjects will be assigned an Investigation identification number by the study site sequentially

starting with 001 upon enrolment into the study. The study site will maintain a master Subject Identification Log.

b. Record keeping and archiving

Archiving will be authorised by the Sponsor following submission of the end of study report. Chief Investigators

are responsible for the secure archiving of essential Investigation documents as per their Trust policy. All essential

documents will be archived for at least 5 years after completion of Investigation. Destruction of essential

documents will require authorisation from the Sponsor.

The Chief Investigator will ensure there are adequate quality and number of monitoring activities conducted

by the study team. This will include adherence to the protocol, procedures for consenting and ensuring

adequate data quality.

The Chief Investigator will inform the sponsor should he/she have concerns which have arisen from

monitoring activities, and/or if there are problems with oversight/monitoring procedures.

An independent data monitoring committee (IDMC) will be set up to deal with patient safety issues related

to this project. The IDMC will comprise of three independent researchers at the Institute of Neurology not

linked to this project.

The data to be monitored by the IDMC will be taken from the CRFs (which will include all AEs and ADEs),

as indicated above.

A.12 Statistical Considerations

**Design** 

A small, well-defined sample of patients with the potential to benefit from the DNI will be recruited. The main

outcome measure is whether the DNI is effective at improving naming impairments. This comparison is within-

subject and is achieved by comparing post-therapy measures to multiple baseline measures. We also compare two

different versions of the therapy in order to answer our secondary question of whether the therapy can be optimised

(a between-groups comparison).

Sample size calculation

Gotcha! sample size is derived from a 5% two sided significance level. This calculation is based on 3-

month follow-up data (change in naming accuracy) taken from Clare et al, 2002. Trained items value

change = 2.55 [SD:2.20]; control items (untrained) value change = 0.91 [SD:1.86] Alpha error = 5%;

Power = 80%. Sample size = 25 in both groups. Expected drop-out rate is 15% so overall we will recruit

44 participants.

Planned recruitment rate

We will begin recruitment prior to the start of the trial and hope to have 50% of patients enrolled by the

time the first patient enters the trial.

Randomisation methods

After Gotcha! participants complete baseline testing (time-point 3) they will be randomised using

minimisation to make sure the groups do not become unbalanced on key baseline variables. This will

determine if they go into the Gotcha! (only) group or Gotcha! maintenance group.

Participants will be randomised on the following variables for Gotcha!: dementia severity (ACEIII) & onset of

diagnosis of dementia.

Multivariate analyses that adjust for all factors used in the minimisation algorithm will be performed as will the

Digital Interventions in Neuro-Rehabilitation: Gotcha! CIP. Version: 6, Date: 15.01.24, IRAS #: 237795


appropriate sensitivity analyses.

Statistical analysis

Behavioural baseline data will be used to ensure that the two groups are not unbalanced on key demographic

variables, including baseline performance during the randomisation procedure. This process of randomisation is

called minimisation (Altman, BMJ 2005).

Data from all time points will be analysed using a repeated-measures ANOVA to determine whether there is an

interaction between time (therapy block vs baseline) and item (trained vs untrained). The effect of the between-

group factor (therapy type) is a secondary outcome measure which will also be analysed using a repeated measure

ANOVA but with this extra factor added in: more formally, a three-way interaction between time (therapy block vs

baseline), item (trained vs untrained) and therapy type (Gotcha! vs Gotcha! maintenance).

Neuroimaging data, collected at three of the time points: Structural magnetic resonance imaging (MRI) data will be

used to identify the lesion location and to aid co-registration of the functional MEG data. Brain structure at the

three time points will be analysed using Voxel-Based Morphometry (Ashburner and Friston 2000) within the

Statistical Parametric Mapping software (SPM12) to identify whether these therapies induce any structure brain

changes over time. We will employ multi- parameter mapping MRI methodology for the structural brain scans

(Callaghan et al, 2014). Brain imaging data (both functioning, structural and MEG) will be analysed using

statistical parametric mapping 12 software (http://fil.ion.ac.uk/sp,). Structural MRI scans will be analysed using

Voxel Based Morphometry (VBM, Ahsbrner & Friston, 2000) to test for therapy-induced changes in brain

structure.

**Missing Data** 

We expect a 15% drop out rate (see sample size correlation above). If the drop out rate is less than 5% then we will

remove these cases and proceed with a per-protocol analysis. For drop out rates over 5% we will assess the impact

of any potential missing data on our study by conducting the following sensitivity analyses:

1) Categorise the missing data – Missing completely at random (MCAR), Missing at random (MAR) or

Missing not at random (MNAR).

If any patients drop out of this study details as to why will be collected from the patient at the time of dropout. The

reasons given will be used to categorise the missing data and justify subsequent handling of the missing data.

2) Handling missing data –

a) MCAR:

In this case the relevant cases will be deleted using listwise or pairwise deletion as appropriate using SPSS.

b) MAR and MNAR:

We will use multiple imputation methods to generate multiple copies of the original dataset by replacing missing values using an appropriate model. Analyse as complete data sets and combine the different parameter estimates

across the data sets to produce a unique point estimate and standard error taking into account the uncertainty of the

imputation process.

3) Sensitivity Analyses

We will compare the results of the full dataset analysis (dataset with imputed values) to those of the complete case

analysis (dataset with observed data only) on a case-by-case basis. To assess the impact of any missing data on the

conclusions of the study.

A.13 Data Management

The handling of all data on the CRFs will be the responsibility of UCL.

It will be the responsibility of the investigator to ensure the accuracy of all data entered in the CRFs. The

delegation log will identify all those personnel with responsibilities for data collection and handling, including

those who have access to the trial database.

We believe that this DNI will be easy to use and that participants will want to do their therapy as the

experience of it being a digital game will be pleasurable. However, therapy is difficult and tiring so in order

to minimise possible distress or frustration, the research team will systematically call the participants if they

are struggling to meet their targets of therapy week by week. This will enable the participant to discuss any

barriers to doing the therapy and researchers can check in with participants to solve any possible, but

unlikely, technical issues.

A13.1 Procedures for data review, database cleaning, and issuing and resolving data queries.

Data entered on the CRFs will be source verified by a sponsor representative trained on the CIP and who has

current GCP training. Data Clarification Forms (DCF) will be issued to the Investigator should a discrepancy be

found between the source and CRF. The Investigator will be required to verify and correct all errors or provide an

explanation for the discrepant data. Sponsor representatives will re-verify the corrected data and mark the

clarification as resolved at the next monitoring visit.

A13.2 Procedures for verification, validation and securing of electronic clinical data systems

All data from the examinations and investigations listed in Appendix A will be transferred to media

provided by the sponsor and collected at the time of CRF collection.

The CI will manage and maintain the study database throughout the Investigation. At the conclusion of the

Investigation, the database will then be locked and data transferred for analysis. A final copy of the database will

be provided to the study site. Where data is transferred electronically, this will be in accordance with the UK Data

Protection Act 1998 as well as Trust Information Governance Policy. There will be a documented record of data

transfer and measures in place for the recovery of original information after transfer.

The database maintained by the CI shall be validated and secured according to the UCL standard operating

procedures. Access to the data shall be limited to sponsor representatives directly involved in the collection,

analysis, maintenance or safety monitoring of the data. Any study data released shall be done according to

the publication policy and in accordance with the UK Data Protection Act 1998.

A13.3 Data retention

Archiving will be authorised by the Sponsor following submission of the end of study report. Chief Investigators

are responsible for the secure archiving of essential Investigation documents and the Investigation database as per

their trust policy. All essential documents will be archived for at least 20 years after completion of Investigation.

Destruction of essential documents will require authorisation from the Sponsor.

A13.4 Clinical quality assurance

The Clinical Investigators will meet monthly, to discuss any issues with data quality and any concerns will be

discussed with the Sponsor.

A13.5 Completion of Case Report Forms

The Principal investigator will be responsible for the timing, accuracy and completeness of a CRF for each

individual subject. All entries are to be made in black ink and are to be legible. All corrections made are to be

completed by placing a single line through the incorrect data and the individual making the correction must initial

and date the correction. Typing correction fluid must not be used. The personal data recorded on all documents will

be regarded as confidential.

The Principal investigator must record the subject's participation in this clinical investigation in the subject's

hospital notes. In addition, the Principal investigator must keep a separate list of all subjects entered into the

clinical investigation showing each subject's name, date of birth and assigned subject number (for identification

purposes). A Subject Identification Log will also be provided in the Investigation Site File to record the subject's

initials and assigned subject number.

All data will be handled in accordance with the UK Data Protection Act 1998.

The CRFs will not bear the subject's name or other personal identifiable data. The subject's initials, date of birth

and trial identification number, will be used for identification.

A13.6 Review and Return of Completed Documentation

The Principal investigator will make the original Case Report Forms available to the Sponsor's designated monitor

at each visit. At the conclusion of the clinical investigation, completed Case Report Forms will be signed by the

Principal investigator, collected (the original left with the Principal investigator) and a copy returned to the

Sponsor.

A13.7 Retention of Documentation

The Principal investigator will retain all copies of the records for a period of 20 years from the discontinuation of

the clinical investigation. In all cases, the Principal investigator must contact the Sponsor prior to disposing of

any records related to the clinical investigation. Included in records to be maintained are signed Clinical

Investigation Plan, copies of the CRFs, signed consent forms, ethics committee approval letters, product

accountability records, correspondence concerning the clinical and any other documents to identify the subjects.

In addition, if the Principal investigator moves/retires, etc., he should provide University College London with

the name and address of the person who will look after and be responsible for the clinical investigation related

records.

Digital Interventions in Neuro-Rehabilitation: Gotcha! CIP. Version: 6, Date: 15.01.24, IRAS #: 237795


A13.8 Training

During the initiation of the investigation site, the sponsor will ensure the investigators and the site study staff are

trained on the device. The investigator is then responsible for ensuring that the investigation staff uses the device

in the same way. All training will be documented in a Site Training Log.

The monitor will also ensure that the investigator and investigation site team have received and understood the

requirements and content of:

\* CIP (Clinical Investigation Plan)

\* IB (Investigators Brochure)

\* The informed consent forms

\* CRFs (Case Report Forms)

\* IFUs (Instructions For Use)

\* All written clinical investigation agreements as appropriate

A.14 Amendments to the CIP

Amendments to this CIP may be necessary to protect the safety of the patients and integrity of the data. In

collaboration with the Investigator(s), the CIP amendments will be documented and submitted for ethical and

regulatory approval (as required) prior to implementation. All changes will be evaluated for impact per sponsor

SOPs. Amendments will be considered implemented after all ethical and regulatory approvals (as required) are

received and all key sponsor and site staff has been trained. This process does not affect the individual clinician's

responsibility to take immediate action if thought necessary to protect the health and interest of individual patients.

A.15 Deviations from clinical investigation plan

A deviation is considered a departure from the conditions and principles of GCP in connection with that

Investigation; or the CIP relating to that Investigation, as amended from time to time.

The Investigator shall not deviate from this CIP except in situations that affect the subject's rights, safety and well-

being, or the scientific integrity of the clinical investigation.

A.15.1 Procedures for recording, reporting and analysing CIP deviations

If possible, prior approval from the sponsor and REC, if appropriate, shall be obtained by the investigator. All

spontaneous CIP deviations shall be recorded and reported to the sponsor as agreed. A deviation log shall be

maintained by the study site. Deviations shall be reported to the REC and the regulatory authorities if required by

national regulations. All deviations will be included, as required in the final study report.

Notification requirements and time frames.

Requests for deviations by the investigator will be responded to within 48 hours of receipt.

Corrective and preventive actions and principal investigator disqualification criteria.

Refer to the Monitoring Plan (as applicable) for corrective and preventative actions and principal investigator

disqualification criteria.

A.15.2 Procedure for reporting any protocol deviations

Any deviation from the protocol that has not been previously approved by the sponsor (JRO at University College

London), must be reported to the sponsor within 2 working days of the deviation occurrence. Any deviations from

the clinical investigation plan that are identified during routine monitoring visits will be reported to the sponsor

(JRO, University College London) within 24 hours of being identified.

A.16 Statements of compliance

The clinical investigation shall be conducted in accordance with the ethical principles of the Declaration of

Helsinki, ISO standard 14155 and all other applicable device and UK regulations.

The clinical investigation shall not commence recruitment until all REC, regulatory (if applicable) and local (NHS

permission) is received. All additional requirements imposed by the REC or regulatory authority will be followed.

A.17 Insurance

University College London holds insurance against claims from participants for injury caused by their participation

in the clinical trial. Participants may be able to claim compensation if they can prove that UCL has been negligent.

However, as this clinical trial is being carried out in a hospital, the hospital continues to have a duty of care to the

participant of the clinical trial. University College London does not accept liability for any breach in the hospital's

duty of care, or any negligence on the part of hospital employees. This applies whether the hospital is an NHS Trust or otherwise.

Participants may also be able to claim compensation for injury caused by participation in this clinical trial without the need to prove negligence on the part of University College London or another party. Participants who sustain injury and wish to make a claim for compensation should do so in writing in the first instance to the Chief Investigator, who will pass the claim to the Sponsor's Insurers, via the Sponsor's office.

Hospitals selected to participate in this clinical trial shall provide clinical negligence insurance cover for harm caused by their employees and a copy of the relevant insurance policy or summary shall be provided to University College London, upon request.

There must also be indemnity arrangements in place, with the manufacturer, to cover the malfunction and breakdown of the device. N/A

### A.18 Adverse events, adverse device effects and device deficiencies

## a-c) Definitions

| Term | Definition |
|---|---|
| Adverse Event (AE) | Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device. Note 1: This definition includes events related to the investigational medical device or the comparator Note 2: This definition includes events related to the procedures involved Note 3: For users or other persons, this definition is restricted to events related to investigational medical devices |
| Adverse Device Effect<br>(ADE) | Adverse Event related to the use of an investigational device. Note 1: This definition includes AEs resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational device Note 2: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device |
| Serious Adverse Event<br>(SAE) | <ul> <li>Any adverse event that:</li> <li>Led to death,</li> <li>Led to serious deterioration in the health of the subject, that either resulted in</li> <li>a life-threatening illness or injury, or</li> <li>a permanent impairment of a body structure or a body function, or</li> <li>in-patient or prolonged hospitialisation, or</li> <li>medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,</li> <li>Led to foetal distress, foetal death or a congenital anomaly or birth defect</li> </ul> |

| Serious Adverse Device Effect (SADE) | An ADE that has resulted in any of the consequences characteristic of an SAE |
|---|---|
| Unanticipated Serious<br>Adverse Device Effect<br>(USADE) | An SADE, which by its nature, incidence, severity or outcome, has not been identified in the current version of the risk analysis report. |
| Device Deficiency (DD) | Inadequately of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Note 1: this includes malfunctions, use errors, and inadequate labeling |

## An adverse event does not include:

- Medical or surgical procedures; the condition that leads to the procedure is an adverse event.
- Pre-existing disease, conditions, or laboratory abnormalities present at the start of the study that do not
  worsen in frequency or intensity.
- Situations where an untoward medical occurrence has not occurred (e.g., hospitalizations for cosmetic or elective surgery or social/convenience admissions);
- The disease being studied or signs/symptoms associated with the disease unless more severe than expected for the subject's condition.

## d) Reporting requirements and timelines

AEs and ADEs are not considered reportable.

| Term | Reporter | Reported to | Reporting Timeline from awareness of the event |
|---|---|---|---|
| Adverse Event (AE) | Investigator | Sponsor | As agreed with sponsor. CI to record fully all AEs. |
| Adverse Device Effect (ADE) | Investigator | Sponsor/Manufacturer | As agreed with sponsor. CI to record fully all ADEs. |

The following events are considered reportable events in accordance with Annex 7, section 2.3.5 and Annex X, section 2.3.5 of DIRECTIVES 90/385/EEC AND 93/42/EEC respectively.

| Term | Reporter | Reported to | Reporting Timeline from awareness of the event |
|---|---|---|---|
| Serious Adverse Event | Investigator | Sponsor | Immediately, but no more than 3 calendar days after becoming aware of the event |
| (SAE)**/ Serious<br>Adverse Device Effect<br>(SADE) | CI | MHRA aic@mhra.gsi.gov.uk | Immediately, but not later than 2* calendar days after awareness *For SAEs which indicate an imminent risk of death, serious injury, or serious illness and |

| | CI | REC | that require prompt remedial action for other patients/subjects, users or other persons All other events immediately but not later than 7 calendar days following date of awareness. N/A |
|---|---|---|---|
| | Investigator | Sponsor | Immediately, but no more than 3 calendar days after becoming aware of the event |
| | CI | MHRA | Immediately, but not later than 2* calendar days after awareness |
| Unanticipated Serious<br>Adverse Device Effect<br>(USADE) | | | *For SAEs which indicate an imminent risk of death, serious injury, or serious illness and that require prompt remedial action for other patients/subjects, users or other persons. All other events immediately but not later than 7 calendar days following date of awareness. |
| | CI | REC | Within 15 days of the chief investigator becoming aware of the event. Only reports of related and unexpected Serious Adverse Events (SAEs) should be submitted to the REC. |

| Term | Reporter | Reported to | Reporting Timeline from awareness of the event |
|---|---|---|---|
| | Investigator | Sponsor | Immediately, no more than 24 hours of becoming aware of the event |
| Device Deficiency<br>(DD) | CI | MHRA | 7 calendar days Only reportable if the event may have led to an SAE if; • suitable action had not taken • intervention had not been made • if circumstances had been less fortunate |
| Urgent Safety<br>Measures | CI | REC | <ul><li>(i) Immediately-By telephone</li><li>(ii) Within 3 days-Notice in writing setting out reasons</li></ul> |

| for the USM and plan for further action |
|-----------------------------------------|

<sup>\*\*</sup> **Note** Planned hospitalisation for a pre-existing condition, or a procedure required by the CIP, without serious deterioration in health, is not considered a serious adverse event

## e) Assessments of adverse events

Each adverse event will be assessed for the following criteria:

## **Severity**

| Category | Definition |
|---|---|
| Mild | The adverse event does not interfere with the subjects daily routine, and does not require intervention; it causes slight discomfort |
| Moderate | The adverse event interferes with some aspects of the subjects routine, or requires intervention, but is not damaging to health; it causes moderate discomfort |
| Severe | The adverse event results in alteration, discomfort or disability which is clearly damaging to health Note: A severity rating of severe does not necessarily categorise the event as an SAE. |

### Seriousness

Seriousness as defined for an SAE in section a) above.

## **Causality**

The assessment of relationship of adverse events to the study procedure and the investigational device will be a clinical decision based on all available information at the time of the completion of the case report form. The following categories will be used to define the causality of the adverse event:

| Category | Definition |
|---|---|
| Yes | There is evidence to suggest a causal relationship, and the influence of other factors is unlikely |
| Possibly | There is some evidence to suggest a causal relationship (e.g. the event occurred within a reasonable time after procedure). However, the influence of other factors may have contributed to the event (e.g. the patient's clinical condition, other concomitant events). |
| No | There is no evidence of any causal relationship. |

## **Expectedness**

| Category | Definition |
|---|---|
| Expected | An adverse event that is consistent with the information about the |

| | device listed in the Investigator Brochure or clearly defined in this CIP. |
|---|---|
| Unexpected | An adverse event that is <u>not consistent</u> with the information about the device listed in the Investigator Brochure |

The reference document to be used to assess expectedness against the intervention is the IB. The CIP will be used as the reference document to assess disease related and/or procedural expected events.

### f) Procedures for recording and reporting Adverse Events and Device Deficiencies

Investigator responsibilities:

All adverse events and SAEs will be recorded in the medical records and CRF following consent.

All serious adverse events will need to be reported to the sponsor on a SAE form (using MEDDEV form 2.7/3) unless stated in the CIP that some expected SAEs will not be reported to the sponsor, with a justification as to why they will not be reported.

For patients on the control arm of an Investigation, SAEs may not have to be reported to the sponsor but will be recorded in the CRF and medical records.

The Chief or Principal Investigator will complete the serious adverse event form and the form will be emailed to the sponsor UCL, within 3 working day of his/her becoming aware of the event. The Chief or Principal Investigator will respond to any SAE queries raised by the sponsor as soon as possible.

The Investigator will report to the MHRA and REC (as applicable) all reportable events within the specified timeframes as per section d above.

All deaths will be reported to the sponsor irrespective of whether the death is related to disease progression, the device, or an unrelated event.

All serious adverse events will be recorded in the medical records and the CRF, and the sponsor's AE log.

All SAEs (except those specified in section d as not requiring reporting to the Sponsor) must be recorded on a serious adverse event (SAE) form. The CI/PI or designated individual will complete the sponsor's SAE form and the form will be preferably emailed to the Sponsor within 5 working days of becoming aware of the event. The Chief or Principal Investigator will respond to any SAE queries raised by the sponsor as soon as possible. Where the event is unexpected and thought to be related to the intervention, this must be reported by the Investigator to the Health Research Authority within 15 days.

Digital Interventions in Neuro-Rehabilitation: Gotcha! CIP. Version: 6, Date: 15.01.24, IRAS #: 237795  All SAEs and UADEs should be reported to the following; Cambridge East REC and the MHRA.

Reporting of all Adverse Events and Device Deficiencies: Investigator and Sponsor responsibilities

Investigator responsibilities shall be as per section d). The sponsor shall keep detailed records of all adverse events

and device deficiencies relating to the clinical Investigation, which are reported to them by the Investigation

investigators. The sponsor shall ensure that all relevant information about a reportable event, which occurs during

the course of this clinical Investigation in the United Kingdom, is reported as soon as possible to the MHRA, and

the relevant ethics committees per their reporting requirements and according to the timelines in section d. Any

additional relevant information should be sent within the same time frame as the initial report. The CI is

responsible for informing the appropriate regulatory authorities, ethics committees and other investigators of any

reportable events that have occurred with the study device in any clinical investigation according to the guidelines

set forth by either the REC of record or regulatory authority in the country where the clinical investigation is taking

place.

**Progress reports** 

Progress reports will be submitted to the REC as per the REC requirements. The chief investigator will prepare the

annual progress reports.

Foreseeable adverse events and anticipated adverse device effects

a) Anticipated adverse events and adverse device effects (ADEs), together with their likely incidence,

mitigation or treatment.

**Adverse events** 

Some progression in dementia is expected however significant changes in the disease profile may also occur.

1) Myocardial infarction.

2) Angina.

3) Peripheral vascular disease.

4) Significant progression of dementia

Digital Interventions in Neuro-Rehabilitation: Gotcha! CIP. Version: 6, Date: 15.01.24, IRAS #: 237795


If any brain abnormality is found on the MRI scans during the study the following procedure will be adhered to: All abnormal structural scans will be shown to a Consultant Neuroradiologist from the National Hospital for Neurology and Neurosurgery, as soon as possible.

Prof Alex Leff, Consultant Neurologist will have responsibility for reporting the finding to the participant's GP and discussing it with the participant as soon as possible.

A record of events will be kept in the research log however they will not be reported to REC and MHRA as they are anticipated events that patients are at risk of due to the nature of the underlying condition being studied. The records of these events will be discussed by the IDMC.

### Adverse device effects and events

Below is a table summarising the anticipated adverse device effects and events.

| Adverse event/effect | Likelihood (low, medium, high) | Mitigation Strategy |
|---|---|---|
| For the G! therapy participants are | Low | Before each G! participant starts |
| required to gather the photo assets | | the trial a member of the research |
| (i.e a picture of someone they | | team will be able to check the |
| wish to remember) and record the | | quality of the audio and photo |
| audio assets (a short 3s audio clip | | assets added to the G! app by each |
| of them saying the person's | | participant. If any are not |
| name). | | acceptable then participants will |
| There is a small risk that poor | | be asked to re-record the assets. |
| quality photo and audio assets | | Additionally participants are given |
| gathered. | | advice at the start of the trial on |
| | | how to take the pictures and |
| | | recordings according to the |
| | | standards needed for the trial. |
| Despite the user and simulation | Medium | During the clinical trial, all bugs |
| testing carried out on | | will be tracked and logged using |
| development. There is still risk of | | the Project Locker bug tracking |
| unanticipated bugs in the software | | tools) and all bugs will be given a |
| that may arise due to differences | | unique reference code, an |
| in patient usage from the | | associated record for that |

| recommended usage. | | reference code is captured, by the |
|---|---|---|
| | | clinical team, detailing what |
| | | caused the bug to occur, each bug |
| | | is then prioritized and a fix is |
| | | implemented (The clinical team |
| | | will have access to the bug |
| | | tracking code reports). Once a bug |
| | | is fixed by the engineering team a |
| | | standard formal automated |
| | | verification test (again a test prior |
| | | approved by the clinical team) is |
| | | run on the compiled software to |
| | | verify that the bug has been fixed. |
| Speech recogniser gives an | Medium | During the trial the performance |
| incorrect binary decision. There is | | of the speech recognizer will be |
| a risk that the speech recognition | | monitored by the research team |
| system may provide incorrect | | via the backend. The speech |
| decisions to patient input i.e false | | recognizer is expected to work at |
| positive or false negative | | 80% accuracy. Thus these types of |
| decisions on a patient's naming | | risks are considered an expected |
| attempt. | | adverse device event and as such, |
| | | a record of these types of events |
| | | will be kept and reviewed by the |
| | | relevant auditing committee and |
| | | the IDMC for the trial. |
| Patient fatigue, headache, | Low | The device can be supported by |
| eyestrain from using the tablet | | the user or can be used with table |
| device during the therapy and | | to prevent any patient fatigue if |
| from prolonged screen time. | | holding the tablet. |
| | | Participants will also be |
| | | encouraged to take regular beaks |
| | | and to avoid prolonged screen |
| | | time. |

A.19 Oversight Committees

**Trial Management Group (TMG)** 

The TMG will include the Chief and Principal Investigators and experts from relevant specialties. The TMG will

be responsible for overseeing the trial. The group will meet at least twice per year and all members will sign a

TMG charter. The TMG will review substantial amendments to the protocol prior to submission to the REC and

MHRA.

**Trial Steering Committee (TSC)** 

As this is not a multicenter trial, the TMG and TSC are one and the same.

**Independent Data Monitoring Committee (IDMC)** 

The role of the IDMC is to provide independent advice on data and safety aspects of the trial. Meetings of the

Committee will be held annually to review the safety data generated by the study or as necessary to address any

issues. Information about adverse events and device effects will be gathered at each of the clinical trial time-points

per patient. If the IDMC deems any adverse event or device effect is excessively high (i.e statistically and

clinically significant) then they can recommend premature closure of the trial.

The IDMC is advisory to the TSC and can recommend premature closure of the trial to the TSC. All IDMC

members will sign an IDMC charter.

A.20 Vulnerable population

a) Description of the vulnerable population.

**Dementia** 

Some people with dementia may be considered vulnerable as they may develop cognitive difficulties.

However, as part of this clinical trial we will not be recruiting anyone with significant cognitive impairment

and therefore on an individual basis may not be considered as vulnerable

There may be some support with travelling to appointments by family members which we will encourage.

b) Description of the specific informed consent process.

### Gotcha!

People with dementia may need more time to process the information and this is why we give a week for them to go through the PIS. Patients who are incapable of providing informed consent (patients without capacity) will not be recruited.

c) Description of the EC's specific responsibility.

N/A

d) Description of what medical care, if any, will be provided for subjects after the clinical investigation has been completed.

N/A

## A.21 Suspension or premature termination of the clinical investigation

Both the Sponsor and the Principal investigator reserve the right to terminate the clinical investigation at any time. Should this be necessary, the procedures will be arranged on an individual basis after review and consultation by both parties. In terminating the clinical investigation, the JRO at University College London and the Principal investigator will assure that adequate consideration is given to the protection of the subject's interests.

## **A21.1 Subject Withdrawals and Discontinuation**

A participant may be withdrawn from the trial whenever continued participation is no longer in the participant's best interests, but the reasons for doing so must be recorded. Reasons for discontinuing the trial may include:

- Subject's rescission of consent.
- Any unexpected adverse device effect which is, in the opinion of the Principal investigator, related to
  the device and will endanger the wellbeing of the subject if the treatment is continued.
- The development of any undercurrent illness(es), infection or condition(s) that might interfere with the Clinical Investigation Plan.
- Any problem deemed by the Principal investigator and/or the JRO at University College London to be sufficient to cause discontinuation.
- Disease progression whilst in the study
- Intercurrent illness
- Patients withdrawing consent

• Persistent non-compliance to protocol requirements.

All subjects discontinued from the clinical investigation due to an unexpected adverse device effect, directly

related to the clinical investigation, will be treated until the effect resolves. The Principal investigator will clearly

document the date and reason(s) for subject withdrawal in his/her CRF and the monitor must be notified.

Subjects who are withdrawn will not be replaced if they have received the investigational device. If possible, any

procedures or assessments planned for the subject on withdrawal from the clinical investigation should be

performed when intention to withdraw the subject is announced.

Subjects who are withdrawn prior to receiving investigational device will be replaced.

A.22 Definition of End of Trial

The expected duration of the trial is 3 years from recruitment of the first participant. The end of the trial (phase 2)

is the date of the last visit of the last participant.

A.23 Publication policy

Yes we plan to publish the findings.

As we are NIHR funded the NIHR need to be sent a draft at the time of submission. The rules are here:

"The NIHR actively encourages the dissemination of research. Investigators and their research teams funded under

an NIHR programme should provide advance notice of research outputs. A copy of the proposed publication

should be sent to the funding programme at the same time as submission for publication or at least 28 days before

the date intended for publication whichever is earlier. Please note this also applies to press releases to be issued by

your host institution, e.g. university, NHS Trust or hospital. (Please see 4.1 on Press Releases)"

https://www.nihr.ac.uk/funding-and-support/documents/funding-for-research-studies/manage-my-

study/outputs-guidance-notes-2.pdf (page 2).

All proposed publications will be discussed with and reviewed by the Sponsor prior to publishing other than those

presented at scientific forums/meetings. Please refer to UCL publication policy.

The results of the study will be reported in the following ways: peer reviewed scientific journals; internal report;

conference presentation; written feedback to research participants.

Please refer to UCL publication policy.

Digital Interventions in Neuro-Rehabilitation: Gotcha! CIP. Version: 6, Date: 15.01.24, IRAS #: 237795


### **Intellectual Property**

All background intellectual property rights (including licences) and know-how used in connection with the study shall remain the property of the party introducing the same and the exercise of such rights for purposes of the study shall not infringe any third party's rights.

All intellectual property rights and know-how in the protocol and in the results arising directly from the study, but excluding all improvements thereto or clinical procedures developed or used by each participating site, shall belong to UCLH. Each participating site agrees that by giving approval to conduct the study at its respective site, it is also agreeing to effectively assign all such intellectual property rights ("IPR") to UCL and to disclose all such know-how to UCL.

Each participating site agrees to, at the request and expense of UCL execute all such documents and do all acts necessary to fully vest the IPR in UCL.

Nothing in this section shall be construed so as to prevent or hinder the participating site from using know-how gained during the performance of the study in the furtherance of its normal activities of providing or commissioning clinical services, teaching and research to the extent that such use does not result in the disclosure or misuse of confidential information or the infringement of an intellectual property right of UCL. This does not permit the disclosure of any of the results of the study, all of which remain confidential.



## A.24 Bibliography

List of the literature and data that are relevant to the trial, and that provide background for the trial. Please ensure the text contains appropriate cross references to this list

- Ashburner, J. and K.J. Friston (2000). "Voxel-based morphometry-the methods". Neuroimage, **11** (6 Pt 1): 805-821.
- Bhogal, S.K., R. Teasell, and M. Speechley (2003). "Intensity of aphasia therapy, impact on recovery". Stroke, **34**(4): 987-93.
- Brady, M.C., H. Kelly, J. Godwin, and P. Enderby (2013). "Speech and language therapy for aphasia following stroke". Cochrane Database of Systematic Reviews, **12**(5).
- Callaghan, J., J. Wells, S. Richardson, H. Holmes, Y. Yichao, S. Walker-Samuel, B. Siow, and M.F. Lythgoe (2014). "Is Your System Calibrated? MRI Gradient System Calibration for Pre-Clinical, High-Resolution Imaging". Plos one: https://doi.org/10.1371/journal.pone.0096568.
- Code, C. and C. Heron (2003). "Services for aphasia, other acquired adult neurogenic communication and swallowing disorders in the United Kingdom, 2000." Disability Rehabilitation 25(21): 1231-1237.
- Clare L., B.A. Wilson, G. Carter, I. Roth, and J.R. Hodges (2002). "Relearning face-name associations in early Alzheimer's disease". Neuropsychology, **16**(4): 538-47.
- Craig P., P. Dieppe, S. Macintyre, S. Michie, I. Nazareth, and M. Petticrew (2008). "Developing and evaluating complex interventions: the new Medical Research Council guidance".

  British Medical Journal, 33(7): a 1655.
- Moss A., and M. Nicholas (2006). "Langauge Rehabilitation in chronic aphasia and time postonset". Stroke, **37**(12): 3043-3051.
- Palmer, R., Enderby, P., Cooper, C., Latimer, N., Julious, S., Paterson, G. & Delaney, A. (2012). Computer therapy compared with usual care for people with long-standing aphasia poststroke: a pilot randomized controlled trial. *Stroke*, *43*(7), 1904-1911.
- Prince, M., M. Knapp, M. Guerchet, M. P. McCrone, M. Prina, A. Comas-Herrea, R. Wittenberg et





al. (2014). "Dementia UK: Update". London: Alzheimer's Society.

Swinburn, K., G. Porter, and D. Howard (2004). "Comprenhensive Aphasia Test". Psychology Press.

Werner, P. (2004). "Beliefs about memory problems and help seeking in elderly persons". Clinical Gerontologist, **27**(4): 19-30.

| Appendix A: | Gotcha! |
|-------------|---------|

| Gotcha! | Baseline<br>1 | Baseline<br>2 | Baseline<br>3 | Treatment | Time-<br>point 4 | Maintenanc<br>e<br>Treatment | Time-<br>point 5 | Time-<br>point 6 | Time-point 7 |
|---|---|---|---|---|---|---|---|---|---|
| Visit # | 1 | 2 | 3 | 6 weeks | | 12<br>weeks | 5 | 6 | 7 |
| Informed Consent | Week 0 | Week 6 | Week 12 | | Week 18 | | Week 30 | Week 42 | Week 54 |
| Medical History | X | | | | | | | | |
| Baseline<br>neuropsych tests | X | | | | | | | | |
| ACE-III | X | | | | | | X | | X |
| PROMS | X | X | X | X | X | X | X | X | |
| Randomisation | | | | | | | | | |
| Brain Scans | | X | X | | X | | | | |
| Device/Treatment | | | | | | | | | |
| Adverse Events review (CRF) | X | X | X | X | X | X | X | X | X |
| Concomitant<br>Medication review | X | | | | | | | | |